CLINICAL TRIAL: NCT01157065
Title: Controlled, Double-Masked, Randomized, Multicenter Study to Evaluate AL-78898A as a Treatment of Exudative AMD
Brief Title: Evaluation of AL-78898A in Exudative Age-Related Macular Degeneration
Acronym: RACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-067
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-04

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Wet AMD; Intravitreal Injection; Macular Degeneration; VEGF treatment
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-78898A (Experimental): Single 50-µL (microliter) intravitreal injection with 12 weeks follow-up
  Interventions: Drug: AL-78898A
- Lucentis (Active Comparator): Single 50-µL (microliter) intravitreal injection with 12 weeks follow-up
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: AL-78898A — Investigational treatment
  Arms: AL-78898A
Drug: Ranibizumab — Anti-vascular endothelial growth factor (VEGF) treatment
  Other Names: LUCENTIS®
  Arms: Lucentis

SUMMARY:
The primary purpose of this study was to demonstrate a biological effect of AL-78898A, as measured by change (reduction) in central subfield (CSF) retinal thickness 4 weeks after a single intravitreal injection, as compared to LUCENTIS.

DETAILED DESCRIPTION:
The study consisted of a Screening Visit (Visit 1), a Day 0 visit (Visit 2), 6 on-therapy visits at Day 1, Weeks 1, 2, 3, 4, and 8 (Visits 3-8), and an Exit Visit at Week 12 (Visit 9). Patients who met all inclusion and exclusion criteria at Visit 1 were randomized in a 3:1 ratio to receive either AL-78898A or LUCENTIS as a single 50-μL injection in the study eye. Additionally, patients received standard therapy for exudative AMD beginning at Week 2/Visit 5 if the patient was not improving per protocol-specified criteria. Beginning at Week 4/Visit 7, patients not improving received standard therapy for exudative AMD at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give informed consent, make the required study visits and follow instructions;
* Newly diagnosed with exudative age-related macular degeneration (AMD);
* Presence of primary juxta- or subfoveal choroidal neovascularization (CNV) secondary to AMD (study eye);
* Best-corrected visual acuity (BCVA) in study eye as specified in protocol;
* No vision-threatening ocular condition other than AMD, in the opinion of the Investigator;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* History or current evidence of macular or retinal disease other than exudative AMD (study eye);
* Any evidence of fibrosis or scarring within the CNV (choroidal neovascularization)lesion (study eye);
* Any evidence of vitreous hemorrhage (study eye);
* History or evidence of surgery (study eye), as specified in protocol;
* Any active systemic infection or ocular/intraocular infection or inflammation in either eye;
* A history or current medical diagnosis of glaucoma or ocular hypertension (study eye), as specified in protocol;
* History or current evidence of a medical condition that may in the opinion of the Investigator preclude the safe administration of test article, adherence to the scheduled study visits, safe participation in the study or affect the results of the study
* History of severe or serious hypersensitivity to any component of the investigational product, reference product or clinically relevant sensitivity to fluorescein dye, as assessed by the Investigator;
* Females of childbearing potential may not participate in the study if pregnant, lactating, or not using adequate birth control methods for the duration of the study;
* Participation in any ocular or non-ocular investigational study within 30 days of screening;
* Has received any approved or investigational therapy for AMD in the study eye with the exception of vitamins;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hosseini, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 14 study centers in the US.
Pre-assignment Details: Of the 99 subjects enrolled, 48 were considered screen failures and were exited from the study prior to randomization. Of the 51 subjects randomized, 2 did not receive treatment. This reporting group includes all randomized subjects who received study medication.
Period: Overall Study
Arm/Group | AL-78898A | Lucentis
Started | 38 | 11
Completed | 38 | 10
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects who received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-78898A | Lucentis | Total
Number analyzed (Participants) | 38 | 11 | 49
Age, Customized [Number; unit: participants]
  18 to 64 years | 3 | 0 | 3
  ≥65 years | 35 | 11 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 4 | 25
  Male | 17 | 7 | 24
Region of Enrollment [Number; unit: participants]
  United States | 38 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction From Baseline in Central Subfield (CSF) Retinal Thickness at Week 4
Description: The thickness of the retina was measured using a non-invasive device that produces cross-sectional and 3D images of the eye. The reduction was calculated by subtracting Week 4 visit value from the Baseline value. A positive number indicates a reduction in thickness compared to baseline, whereas a negative number indicates an increase in thickness. An increase in thickness as compared to baseline may indicate a progression of the underlying disease.
Time Frame: Week 4
Population: All patients who received study medication, completed at least one scheduled post-injection study visit, and did not receive standard therapy prior to Week 4 assessment
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | AL-78898A | Lucentis
Number analyzed (Participants) | 24 | 10
microns
  Baseline | 514.2 (158) | 551.8 (119.0)
  Week 4 | -12.1 (87.2) | 199.9 (139.6)

2. Primary Outcome: Incidence of Events of Special Interest (ESI)
Description: An ESI was a protocol-specified event of scientific and medical concern specific to the Sponsor's product or program where ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. These adverse events could have been serious or nonserious and may have required further investigation in order to characterize and understand.
Time Frame: Up to Day 30
Population: Intent-to-treat (ITT): All patients who received study medication and completed at least one scheduled post-injection study visit
Measure: Number; unit: events
Arm/Group | AL-78898A | Lucentis
Number analyzed (Participants) | 38 | 11
events | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. This reporting group includes all randomized subjects who received study medication.
Description: An adverse event was defined as any untoward medical occurrence in a patient who was administered a study treatment regardless of whether or not the event had a causal relationship with the treatment. Adverse events were obtained as solicited comments from the study patients and as observations by the Investigator as outlined in the study protocol.
Arm/Group | AL-78898A | Lucentis
Serious Adverse Events (participants affected / at risk) | 5/38 | 1/11
Other Adverse Events (participants affected / at risk) | 14/38 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL-78898A (N=38) | Lucentis (N=11)
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 — Not related
Fall (Injury, poisoning and procedural complications) | 1 | 0 — Not related
Syncope (Nervous system disorders) | 1 | 0 — Not related
Transient ischaemic attack (Nervous system disorders) | 2 | 0 — Not related
Death (General disorders) | 0 | 1 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AL-78898A (N=38) | Lucentis (N=11)
Conjunctival haemorrhage (Eye disorders) | 7 | 1
Eye irritation (Eye disorders) | 3 | 0
Vitreous floaters (Eye disorders) | 3 | 0
Retinal pigment epithelial tear (Eye disorders) | 2 | 0
Eye pruritis (Eye disorders) | 0 | 1
Lens disorder (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.